CLINICAL TRIAL: NCT00906061
Title: Phase II Study of Biweekly Gemcitabine and Docetaxel as First Line Therapy for Advanced Non-Small Cell Lung Cancer Patients With ECOG PS 2
Brief Title: Biweekly Gemcitabine and Docetaxel as First Line Therapy for Advanced Non-Small Cell Lung Cancer (NSCLC) Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Arnau de Vilanova (Other)
Responsible Party: Vicente Alberola Candel, ASOCIACIÓN TERAPEUTICA EN HEMATOLOGÍA Y ONCOLOGÍA MÉDICAS H. ARNAU DE VILANOVA
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPNM-PS2-07
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Small Cell; Lung Neoplasms; Docetaxel; Gemcitabine; ECOG 2
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Small Cell; Lung Neoplasms | interventions — Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine and Docetaxel (Experimental): Patients received biweekly docetaxel 50 mg/m2 iv, Gemcitabine 2000 mg/m2 iv days 1 and 14.
  Interventions: Drug: Gemcitabine and Docetaxel

INTERVENTIONS:
Drug: Gemcitabine and Docetaxel — Docetaxel 50 mg/m2, IV, and Gemcitabine 2000 mg/m2, IV, on day 1 and 14 of each 28 day cycle. Number of Cycles: 6

SUMMARY:
There is little information of Eastern Cooperative Oncology Group (ECOG) performance status (PS) 2 patients analyzed in the clinical trials. The rate of patients recruited into Treatment Chemotherapy as 1st Line in Advanced NSCLC clinical trials is less than 20 percent.

This low rate makes the investigators think about the possibility of a bias selection, due to the existence of this exclusion criteria that do not permit to include patients with deteriorated performance status.

In these types of patients, the toxicity is an important issue to decide the therapeutic strategy. Gemcitabine and Docetaxel combination is very interesting because they have a different toxicity profile. This combination has demonstrated activity in several types of tumours, as breast cancer, sarcoma and lung cancer.

The strategy performed in this study is biweekly combination of Gemcitabine and Docetaxel; activity and dose intensity will be the same, but toxicity will be significantly low.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced NSCLC.
* Stage III with pleural effusion and stage IV.
* Patients with ECOG PS 2.
* Patients must have at least one measurable lesion, no previously irradiated.
* Life expectancy of at least 12 weeks.
* Adequate organ function according to the following criteria:

  * Bone marrow: ANC => 2.0x10(9)cells/L; Platelet count => 100x10(9)cells/L; Hemoglobin => 10 g/dL.
  * Liver function: Bilirubin <= 1.5 X ULN; Alkaline phosphatase <= 5 x ULN; AST and ALT <= 1.5 x ULN.
  * Renal function:serum creatinine <= 2mg/dL.

Exclusion Criteria:

* Prior systemic chemotherapy for advanced disease.
* Prior radiotherapy for NSCLC.
* Patients with symptomatic brain metastases.
* No measurable bone metastases or malignant pleural effusion as only measurable lesion.
* History of prior malignancies, except curatively treated in situ carcinoma of the cervix or other cancer curatively treated and with no evidence of disease for at least five years.
* History of hypersensitivity reaction study drugs.
* Pregnant or lactating women (women of childbearing potential must use adequate contraception).
* Concurrent treatment with other experimental drugs.
* Current peripheral neuropathy NCI grade 2.
* Participation in clinical trials within 30 days of study entry.
* Major surgery, open biopsy or traumatic lesion 28 days before to study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Overall response rate = sum of complete and partial tumour responses divided by the number of included patients | 2 and 4 months

SECONDARY OUTCOMES:
Overall survival | Time from study entry to death from any cause
Toxicity | Biweekly
Duration of response | time from first response (CR or PR) to tumor progression
Time to progression | time from study entry to observed tumor progression or death due to progression disease
Measurement of quality of life | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Juan, Doctor, Study Director — Hospital Arnau de Vilanova de Valencia; Alfredo Sanchez, Doctor, Principal Investigator — Hospital Provincial de Castellón; José Muñoz, Doctor, Principal Investigator — H. Universitario Dr. Peset; Sonia Maciá, Doctor, Principal Investigator — Hospital General de Elda; Vicente Giner, Doctor, Principal Investigator — Hospital de Sagunto; José Gomez, Doctor, Principal Investigator — Hospital Universitario La Fe; Gaspar Esquerdo, Doctor, Principal Investigator — Hospital Clínica de Benidorm; Antonio López, Doctor, Principal Investigator — Hospital San Juan de Alicante; Francisco Aparisi, Doctor, Principal Investigator — Hospital Virgen de los Lirios; Miguel A. Muñoz, Doctor, Principal Investigator — Instituto Valenciano de Oncología; Juan L. Martí, Doctor, Principal Investigator — Hospital Universitario de Alicante; Silvia Catot, Doctor, Principal Investigator — Hospital Althaia, Xarxa Asistencial de Manresa
Locations (12):
- Spain (12):
  - Hospital Virgen de los Lirios, Alcoy, Alicante
  - Hospital Universitario de Alicante, Alicante, Alicante
  - Hospital San Juan de Alicante, Alicante, Alicante
  - Hospital Clínica de Benidorm, Benidorm, Alicante
  - Hospital General de Elda, Elda, Alicante
  - Hospital Althaia, Xarxa Asistencial de Manresa, Manresa, Barcelona
  - Hospital Provincial de Castellón, Castellon, Castellón
  - Hospital de Sagunto, Sagunto, Valencia
  - Hospital Universitario La Fe, Valencia, Valencia
  - Instituto Valenciano de Oncología, Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia, Valencia